CLINICAL TRIAL: NCT03372655
Title: Prognstic Factors Affecting Duchenne Muscular Dystrophy
Brief Title: Prognostic Factors Affecting Duchenne Muscular Dystrophy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nehal Refaat Mohammed, Sponsor investigator, Assiut University
Other Study IDs: PFADMD
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determination of prognostic factors affecting ambulation of duchenne muscular dystrophy

DETAILED DESCRIPTION:
Duchenne muscular dystrophy is the most common herditary muscular disease , it lead to loss of ambulation in early teenageers . It lead to early death at the mean age of 19 years

ELIGIBILITY:
Inclusion Criteria:

* any male pt diagnosed as duchenne muscular dystrophy by typical clinical picture &shooting serum CPK level &EMG study or biopsy & age 10 to 18yrs old

Exclusion Criteria:

* female patient ' age below 10 yrs old or above 18 yrs old .patient with autoimmune disease or malignancy

Ages: 10 Years to 18 Years | Sex: Male
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Male patient diagnosed as duchenne muscular dystrophy by typical clinical picture&shooting serum CPK level & EMG study or biopsy
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Ten meter walking test | 2018 - 2019
  Questionnaire

SECONDARY OUTCOMES:
Muscle strenght | 2018- 2019
  Questionnaire